CLINICAL TRIAL: NCT02243683
Title: A Randomized, Placebo Controlled, Double Blind, Dose Escalating, Crossover, Safety and Pharmacokinetic Study of AX-024.HCl in Healthy Male Subjects
Brief Title: Safety Study of Immune System Modulator for Autoimmune Diseases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Artax Biopharma Inc (Industry)
Collaborators: Simbec Research (Industry); ORION Clinical Services (Industry); Packaging Coordinators Inc (Other); Centro de Biología Molecular Severo Ochoa, Spain (CBMSO) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: AX-024-1.01
Record Dates: First submitted 2014-09-16; First posted 2014-09-18 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Cohort A (Experimental): Single ascending oral administrations of AX-024.HCl (hydrochloride) and matching placebo
  Interventions: Drug: AX-024.HCl; Other: Placebo
- Cohort B (Experimental): Single ascending oral administrations of AX-024.HCl (hydrochloride) and matching placebo
  Interventions: Drug: AX-024.HCl; Other: Placebo

INTERVENTIONS:
Drug: AX-024.HCl
Other: Placebo

SUMMARY:
The purpose of this study is to determine the toxicity, tolerability and safety of single ascending doses of AX-024.HCl in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a body mass index (BMI) of 18 - 35 kg/m2, inclusive. BMI = Body weight (kg) / [Height (m)]2.
* In good health as determined by medical history, physical examination, and clinical judgment of the investigator
* Subject with no history of autoimmune disease or cardiac disease
* Subjects must be available to complete the study (including follow-up visit).
* Subjects must satisfy a medical examiner about their fitness to participate in the study.
* Subjects must provide written informed consent to participate in the study.

Exclusion Criteria:

* A clinically significant history of gastrointestinal disorder likely to influence drug absorption.
* Receipt of regular medication within 21 days of the first dose that may have an impact on the safety and objectives of the study (at the Investigator's discretion).
* Evidence of renal, hepatic, central nervous system, respiratory, cardiovascular or metabolic dysfunction.
* Subjects who are smokers, or ex-smokers who have smoked in the last 3 months (determined by negative urine cotinine at screening visit).
* A clinically significant history of hypersensitivity (anaphylaxis, angioedema) to any drug.
* A clinically significant history of drug or alcohol abuse.
* Participation in a New Chemical Entity clinical study within the previous 4 months or a marketed drug clinical study within the previous 3 months. (N.B. washout period between studies is defined as the period of time elapsed between the last dose of the previous study and the first dose of the next study).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | Over a 72 hours period and 7 days after last dose

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve | Over a 72 hours period post dose

CONTACTS AND LOCATIONS:
Overall Officials: Girish Sharma, MBBS, Principal Investigator — Simbec Research
Locations (1):
- Simbec Research Ltd, Merthyr Tydfil, Cardiff Road, United Kingdom